CLINICAL TRIAL: NCT01374945
Title: Clearpath Miniprep Colonoscopy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn for business reasons
Sponsor: EasyGlide (Industry)
Other Study IDs: EasyGlide-CL-001
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC preparation and colonoscopy (No Intervention)
- Miniprep and Clearpath (Experimental)
  Interventions: Device: Clearpath Lower GI

INTERVENTIONS:
Device: Clearpath Lower GI — Clearpath device for cleaning of colon by irrigation and evacuation
  Arms: Miniprep and Clearpath

SUMMARY:
Use of Clearpath to facilitate successful completion of colonoscopy procedures with sub-optimal preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18-70 years
2. Scheduled for colonoscopy
3. Providing informed consent

Exclusion Criteria:

1. Known large polyps (> 2 cm) for polypectomy
2. Inflammatory Bowel Disease (IBD)
3. Previous colonic surgery
4. Known or suspected stricture
5. Significant co morbidity
6. Significant diverticular disease
7. Contraindicated to receive oral Sodium Picosulfate solution

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)